CLINICAL TRIAL: NCT00179868
Title: C-Reactive Protein As a Predictor of Major Transplant Complications in Pediatric Stem Cell Transplant Patients
Brief Title: C-Reactive Protein as a Predictor of Stem Cell Transplant Complications
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: SCT 0403 CRP
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Leukemia; Stem Cell Transplantation
Keywords: cancer; leukemia; stem cell transplant; complications
MeSH Terms: conditions — Neoplasms; Leukemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: C-Reactive Protein levels — Each patient enrolled in the study will have a serum quantitative c-reactive protein (crp) level drawn on the day of transplant, day 7 of transplant, and twice weekly after that until recovery of neutrophil count (approximately 20-25 days). Patients will be followed for 100 days post-transplant for the development of the following complications:
  1. Sepsis- defined as fever, positive blood culture, need for fluid resuscitation and/or pressor support.
  2. Acute GVHD > grade II defined according to the Seattle criteria
  3. VOD- defined according to the modified Seattle criteria

SUMMARY:
The purpose of this study is to determine if C-Reactive Protein levels are predictive for complications post transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 20 years
* Patient undergoing a stem cell transplant (allogeneic, syngeneic, or autologous) at Childrens' Memorial Hospital
* IRB approved informed consent (and assent for children age 12-17)

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children undergoing a stem cell transplant
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2003-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To determine whether quantitative c-reactive protein measurements can predict major morbidity and mortality in pediatric stem cell transplant patients. | To day +100 post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Morris Kletzel, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Children's Memorial Hospital, Chicago, Illinois, United States